CLINICAL TRIAL: NCT04703023
Title: Vergleich Der Wasseraufnahmefähigkeit Und Zusammensetzung Von Bronchialflüssigkeiten Von Gesunden Und Patienten Mit Chronisch Obstruktiver Bronchitis (COPD)
Brief Title: Comparison of Water Sorption Capacity and the Composition of Bronchial Fluids of Healthy Persons and Patients With Chronic Obstructive Bronchitis (COPD)
Status: Completed | Type: Observational
Sponsor: Georg Nilius, Prof DR med (Industry)
Responsible Party: Sponsor-Investigator, Georg Nilius, Prof DR med, Clinical Director, Institut für Pneumologie Hagen Ambrock eV
Organization: Institut für Pneumologie Hagen Ambrock eV (Industry)
Other Study IDs: MUCUS2020
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: COPD; Healthy
Keywords: mucociliary clearance; mucus; sorption of water
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD: Secretions are collected from Bronchoscopy in clinical routine in COPD patients
- lung healthy: Secretions are collected from Removal of endotracheal tubes after elective surgery in lung healthy patients

SUMMARY:
Pilot basic research study on the properties of bronchial mucus. Examination of the sorption and desorption properties, mucin concentration, and structure of the mucus from healthy airways compared to patients with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Mucus, of the correct composition, maintains airway hydration and protects the airway from inhaled particles through mucociliary transport. In chronic inflammatory airway diseases such as COPD or cystic fibrosis, infectious agents, inflammatory cells and products of inflammation such as DNA, increase mucus viscosity which results in decreased mucociliary clearance of inhaled particles, increasing the likelihood of respiratory infections. This pilot study is planned as basic research on the properties of bronchial mucus.

Water isotherms and efficient water activity (sorption and desorption) of the collected samples are examined in defined temperature and humidity settings using DVS Intrinsic (Dynamic Vapour Sorption System, Surface Measurement Systems, London, UK). Findings will provide insights into possible treatment programs targeted at altering specific mucus components.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* COPD or other disease requiring bronchoscopy or elective surgery
* Signed informed consent form

Exclusion Criteria:

* Not able to consent
* Linguistic, cognitive, or other obstacles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are hospitalized in the Kliniken Essen Mitte
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Sorption | 5 days
  Maximum water sorption per degree of saturation in percent of the dry mass weight of the mucus samples

CONTACTS AND LOCATIONS:
Locations (1):
- Kliniken Essen-Mitte, Evang. Huyssens-Stiftung/Knappschaft gGmbH, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No